CLINICAL TRIAL: NCT06926556
Title: Different Microlenses Array for Controlling Myopia Progression in Children and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: QX-2024-A-003
Record Dates: First submitted 2024-09-28; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Myopia Progressing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- H.M.E.C，High Precision Micro Encircle (Experimental)
  Interventions: Device: Defocus microlenses
- H. A. L. T, highly aspheric lenslet technology (Active Comparator)

INTERVENTIONS:
Device: Defocus microlenses — Different microlenses array (H.M.E.C，High Precision Micro Encircle and H.A.L.T, highly aspheric lenslet technology) for controlling myopia progression in children and adolescents.
  Arms: H.M.E.C，High Precision Micro Encircle

SUMMARY:
This study aims to evaluate the effectiveness of lenses with different defocused microlens array in controlling the progression of myopia in children and adolescents, and to explore the feasibility of effective defocus microlens design, and apply personalized defocus frame lenses for myopia prevention and control.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 6-14 years old;
2. After using 1% cyclohexanone hydrochloride eye drops (Saifeijie) for ciliary muscle paralysis, binocular spherical power were within -0.50D~-4.00D, binocular cylinder power ≤ 1.50D, the anisometropia is less than 1.50D, and the best corrected visual acuity was above 5.0;
3. Within 30 days, the myopia prevention and control methods such as multifocal glasses, orthokeratology, defocusing flexible glasses, progressive glasses, atropine eye drops, red light and acupuncture and moxibustion treatment were not used;
4. The subject has a willingness to receive treatment and an informed consent form is signed by their legal guardian.

Exclusion Criteria:

1. Diagnosed constant strabismus;
2. Diagnosed pathological myopia;
3. Other congenital eye diseases;
4. Researchers believe that the patients have other reasons that are not suitable for inclusion in the project.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 134 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Subjective refraction equivalent spherical | 2 years

SECONDARY OUTCOMES:
Axial length | 2 years

OTHER OUTCOMES:
Other biological parameters | 2 years
  amplitude of accommodation, anterior chamber depth, corneal curvature, white to white distance, central corneal thickness, lens thickness ,pupil size, multispectral refraction topography, choroidal thickness, objective visual quality, wavefront aberration, contrast sensitivity, and strabismus (mahalanobis bar method).
Best corrected visual acuity | 2 years
questionnaires of daily eye habits and wearing time of subjects collected | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Eye Diseases Prevention &Treatment Center/ Shanghai Eye Hospital, School of Medicine, Tongji University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided